CLINICAL TRIAL: NCT02083484
Title: Expanded Access of MK-3475 in Metastatic Melanoma Patients With Limited to No Treatment Options
Brief Title: Program for Pembrolizumab (MK-3475) in Participants With Metastatic Melanoma Who Have Failed Standard of Care Therapy Including Ipilimumab (MK-3475-030)
Status: No longer available | Type: Expanded Access
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 3475-030
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Each participant will receive pembrolizumab every 3 weeks for up to 2 years or until confirmed radiographic disease progression, unacceptable toxicity, confirmed positive pregnancy test, withdrawal of consent, or pembrolizumab approval in the participant's country.

SUMMARY:
This is an expanded access program (EAP) for participants who have progressed after prior systemic therapy including ipilimumab, and V-raf murine sarcoma viral oncogene homolog B1 (BRAF) inhibitor or mitogen-activated protein kinase (MEK) enzyme inhibitor when indicated. Participants cannot be eligible for or have participated in any pembrolizumab (MK-3475) clinical trial with the exception of a participant enrolled in the pembrolizumab protocol MK-3475-006 who received treatment on the ipilimumab treatment arm and progressed; such participants will be eligible to participate in the EAP, regardless of prior treatment with a BRAF/MEK inhibitor, as long as all other eligibility criteria for MK-3475-030 are met.

DETAILED DESCRIPTION:
Pembrolizumab has been approved by the U.S. Food and Drug Administration for the treatment of patients with unresectable metastatic melanoma and disease progression following ipilimumab and if BRAF V600 mutation positive, a BRAF inhibitor. The Expanded Access Program (EAP) for this medicine in the U.S. is closed. The EAP will continue outside the U.S.

ELIGIBILITY:
Inclusion criteria:

* Unresectable (Stage III) or metastatic melanoma
* Failed or progressed on standard of care systemic therapy including ipilimumab (with the exception of a participant with progressive disease while on the ipilimumab arm of MK-3475-006, regardless of prior treatment with a BRAF/MEK inhibitor, as long as all other eligibility criteria for this study are met)
* Willing to sign Informed Consent
* Eastern Cooperative Oncology Group Performance status of 0 or 1
* Female participants of childbearing potential must be willing to use adequate contraception or be surgically sterile, or abstain from heterosexual activity starting with the first dose of treatment through at least 120 days after the last dose of pembrolizumab
* Male participants must agree to use an adequate method of contraception starting with the first dose of treatment through 120 days after the last dose of pembrolizumab
* Adequate organ function

Exclusion criteria:

* Eligible for an accessible pembrolizumab clinical study or previously participated in a pembrolizumab clinical study (with the exception of a participant with progressive disease while on the ipilimumab arm of MK-3475-006)
* Eligible for treatment with a marketed BRAF inhibitor or MEK inhibitor (with the exception of a participant with progressive disease while on the ipilimumab arm of MK-3475-006, regardless of prior treatment with a BRAF/MEK inhibitor, as long as all other eligibility criteria for this study are met)
* Not recovered to Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or better due to prior chemotherapy, radioactive, or biological cancer therapy (including monoclonal antibodies)
* Not recovered from minor or major surgery and less than 4 weeks from major surgery
* History of life-threatening or severe immune-related adverse events on treatment with another immunotherapy
* Expected to require any other form of systemic antineoplastic therapy while receiving pembrolizumab
* History of clinically severe autoimmune disease (e.g., requires chronic immunosuppressive therapy)
* History of pneumonitis, organ transplant, human immunodeficiency virus (HIV), active hepatitis B or hepatitis C
* Active central nervous system metastases, carcinomatous meningitis, untreated brain metastases
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of treatment with pembrolizumab
* Active infection requiring systemic therapy

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Kottschade LA, McWilliams RR, Markovic SN, Block MS, Villasboas Bisneto J, Pham AQ, Esplin BL, Dronca RS. The use of pembrolizumab for the treatment of metastatic uveal melanoma. Melanoma Res. 2016 Jun;26(3):300-3. doi: 10.1097/CMR.0000000000000242. PMID 26848796
- [Result] Bender C, Dimitrakopoulou-Strauss A, Enk A, Hassel JC. Safety of the PD-1 antibody pembrolizumab in patients with high-grade adverse events under ipilimumab treatment. Ann Oncol. 2016 Jul;27(7):1353-4. doi: 10.1093/annonc/mdw128. Epub 2016 Mar 6. No abstract available. PMID 26951629
- [Result] Gangadhar TC, Hwu WJ, Postow MA, Hamid O, Daud A, Dronca R, Joseph R, O'Day SJ, Hodi FS, Pavlick AC, Kluger H, Oxborough RP, Yang A, Gazdoiu M, Kush DA, Ebbinghaus S, Salama AKS. Efficacy and Safety of Pembrolizumab in Patients Enrolled in KEYNOTE-030 in the United States: An Expanded Access Program. J Immunother. 2017 Nov/Dec;40(9):334-340. doi: 10.1097/CJI.0000000000000186. PMID 29028788